CLINICAL TRIAL: NCT02485145
Title: The Analgesic Activity of a Topical Formulation in Patients With Osteoarthritis of the Hands
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Transdermal Therapeutics, Inc. (Industry)
Collaborators: Albert Einstein College of Medicine (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 54321
Record Dates: First submitted 2015-06-17; First posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis of the Hands
Keywords: Topical; Hand osteoarthritis
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A/B (Experimental): In this crossover trial, the A/B group will receive the test product (A) and then the placebo (B). The topical product contains the following: Diclofenac 3%, Baclofen 2%, Orphenadrine Citrate 5% and Bupivacaine 2% in a VersaPro cream, while the placebo is the VersaPro cream alone. Participants will use the test product for 7 days, applying the topical product to the hands twice a day. There will be a 7 day washout period, and then participants will be given the placebo cream, which will be used for 7 days, applying the topical placebo to the hands twice a day.
  Interventions: Drug: A/B; Drug: Placebo
- B/A (Experimental): In this crossover trial, the B/A group will receive the placebo (B) and then the test product (A). The product contains the following: Diclofenac 3%, Baclofen 2%, Orphenadrine Citrate 5% and Bupivacaine 2% in a VersaPro cream, while the placebo is the VersaPro cream alone. Participants will use the placebo product for 7 days, applying the placebo product to the hands twice a day. There will be a 7 day washout period, and then participants will be given the test cream, which will be used for 7 days, applying the topical product to the hands twice a day.
  Interventions: Drug: Placebo; Drug: B/A

INTERVENTIONS:
Drug: A/B — This arm uses the test product first, which consists of Diclofenac 3%, Baclofen 2%, Orphenadrine 5%, and Bupivacaine 2% in a VersaPro cream. This is the A arm. The B arm is the second arm, and consists of the VersaPro cream alone.
  Other Names: Diclofenac 3%; Baclofen 2%; Orphenadrine 5%; Bupivacaine 2%; VersaPro cream
  Arms: A/B
Drug: Placebo — The placebo, which consists of the VersaPro cream, will be utilized in the study.
  Other Names: VersaPro cream
Drug: B/A — This arm uses the placebo product first, which consists of the VersaPro cream alone. This is the B arm. The A arm is the second arm, which consists of the test product which consists of Diclofenac 3%, Baclofen 2%, Orphenadrine 5%, and Bupivacaine 2% in a VersaPro cream. This is the A arm.
  Other Names: Diclofenac 3%; Baclofen 2%; Orphenadrine 5%; Bupivacaine 2%; VersaPro cream
  Arms: B/A

SUMMARY:
Osteoarthritis (OA) affects over 30 million people in the United States and represents our nation's leading cause of disability. Data for the years between 1996-2005, indicate that OA raised overall health care costs by $185.5 billion annually. Largely as a consequence of this disease, the number of patients undergoing joint replacement surgery will quadruple over the next 17 years. Importantly, several recent studies have demonstrated that OA is an independent risk factor for cardiovascular disease . Presently investigators have no medications that alter the natural history of OA. Weight control, exercise and some physical therapy measures are the only interventions short of total joint replacement that alter the course of this disease. To make matters worse, investigators have experienced only setbacks in use of medications aimed at symptom control. Recognition of toxicities of non-steroidal anti-inflammatory drugs (NSAIDs) and narcotic-based analgesics has narrowed the presently available armamentarium for pain control in OA . Clearly OA is a major factor that demands better solutions as the health care system is redesigned.

OA involving the hands represents a major part of the overall burden of this disease. In radiographic surveys about a quarter of the total US population has changes consistent with OA involving the hands. Among the elderly, radiographic hand OA has been found in over half of such individuals and as many as a quarter of them suffer from pain and functional incapacitation. The joints affected typically are the first carpometacarpal (CMC-1) joint, the distal interphalangeal (DIP) joints, and the proximal interphalangeal (PIP) joints . Therapeutic options include acetaminophen, nonsteroidal anti-inflammatory drugs (NSAIDs), and a variety of physical measures such as physical therapy, bracing, and heat and cold applications. To achieve some symptomatic benefit while limiting systemic toxicity, topical therapies have been developed which either act as counter irritants, seek to reduce substance P (capsaicin), or to deliver an NSAID locally through the skin. The leading example of the latter is Diclofenac sodium gel which was shown to reduce pain intensity and improve hand function in a double blind controlled trial. However none of these measures have proven sufficiently effective to meet patient needs. Topical polytherapy will be employed in this study to see if it will be effective against the pain of OA.

DETAILED DESCRIPTION:
A potentially more effective approach is to provide a combination of analgesic and anti-inflammatory agents through a topical delivery system. In the present study compounds with anti-inflammatory and analgesic properties will be combined in a vehicle that promotes penetration of molecules through the skin to deeper underlying tissues such as the joint capsule at articulations in the hands. The vehicle consists of Versapro cream base (a formulation of Medisca, Inc. that contains Vitamin E and Aloe Vera, along with other ingredients that are proprietary), Tranilast powder, Pentoxifylline USP powder, Cetyl Myristoleate 40% wax, liquid Pentylene Glycol, liquid Dimethyl Sulfoxide (DMSO) USP, liquid Propylene Glycol USP, liquid Ethoxy Diglycol reagent, liquid Ethyl Alcohol 190 proof USP. These are all inert ingredients, i.e. they only promote penetration of molecules through the skin. A mixture of the following compounds will be incorporated into this vehicle as the active test medication:

Diclofenac 3% - an NSAID. FDA pregnancy category C for the first 30 weeks, then category D.

Baclofen 2% - an agonist for the GABAB receptors. FDA pregnancy category C.

Orphenadrine 5% - an anticholinergic drug of the ethanolamine antihistamine class. FDA pregnancy category C.

Bupivacaine 2% - a local anesthetic that binds voltage-gated sodium channels and blocks sodium influx into nerve cells preventing depolarization. FDA pregnancy category C.

Due to the FDA pregnancy categories for the drugs used in this study, pregnancy is an exclusion criteria.

The control medication: The vehicle alone will serve as the control compound.

ELIGIBILITY:
Inclusion Criteria:

* OA in at least one hand as defined by ACR Criteria (nodal enlargement in two or more of 10 defined joints, CMC-1, MCP=1, PIPs and DIPs).
* Hand pain duration greater than one year.
* History of NSAID use for hand pain on at least one occasion during the last year.
* Age 40 to 79 years.
* Ability to understand the English language and to comprehend written material at the 5th grade level.

Exclusion Criteria:

* History of psoriasis
* Other painful rheumatic disease, measured by a blood draw that will test for RF factor and ESR.
* Rheumatoid arthritis, as measured by hand x-rays.
* Any diagnosis of fibromyalgia or neurovascular disease.
* Presence of Raynaud's disease.
* -Presence of Raynaud's disease.
* Presence of any peripheral neuropathy.
* Presence of cervical radiculopathy.
* Pregnancy in females (pregnancy test will be administered at intake to females of reproductive capability and their method of birth control recorded.)
* Persons under age 40. Insufficient data are available in adults to judge potential risk in children.
* Those who are not capable of providing informed consent.
* Known allergy to analgesic drugs and the drugs used in this study.
* Those who do not comprehend English. As this is a short-term Pilot study, the potential benefits to the participants is currently unknown. Based upon this knowledge, we believe we are exempt from the requirement to translate the informed consent form into Spanish.
* Those with renal and/or gastrointestinal impairments, i.e. with a creatinine level of 2 and GFS level 4.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
100 mm Visual Analog Scale | Participants will be followed for the 28 days of the study length, with the study measure being given at study day 7, study day 14, study day 21 and study day 28.
  Measurement of OA pain intensity
Australia/Canadian Osteoarthritis Index | Participants will be followed for the 28 days of the study length, with the study measure being given at study day 7, study day 14, study day 21 and study day 28.
  Measurement of osteoarthritis hand function
100 mm Visual Analog Scale | Participants will be followed for the 28 days of the study length, with the study measure being given at study day 7, study day 14, study day 21 and study day 28.
  Global rating of disease activity
Composite Pharmacokinetics | Blood will be drawn at study day 7, study day 14, study day 21, and study day 28
  Participants will be followed for the 28 days of the study length, with the pharmacokinetics being tested at study day 7, study day 14, study day 21 and study day 28 to see the systemic absorption of each of the study drugs. Each drug (Diclofenac, Baclofen, Orphenadrine and Bupivacaine) will be tested for Peak Plasma Concentration (C max) and the area under the plasma concentration versus time curve (AUC).

SECONDARY OUTCOMES:
Use of rescue medication | The entire 28 day study
  Acetaminophen up to 4 grams daily.

CONTACTS AND LOCATIONS:
Overall Officials: John Hardin, M.D., Principal Investigator — Albert Einstein College of Medicine - Yeshiva University and Montefiore Medical Center